CLINICAL TRIAL: NCT06290986
Title: Pyrocardan® Implant Arthroplasty or LRTI for Trapeziometacarpal Osteoarthritis - A Randomized Controlled Trial
Brief Title: Pyrocardan® Implant Arthroplasty or LRTI for Trapeziometacarpal Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Jens Joergsholm, Principal Investigator, PhD student, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pyrocardan® RCT
Record Dates: First submitted 2024-02-14; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: CMC-1 Osteoarthritis; Trapeziometacarpal Osteoarthritis
Keywords: Hand Osteoarthritis; Pyrocardan; CMC-1; Trapeziometacarpal Osteoarthritis; Osteoarthritis; Joint Diseases
MeSH Terms: conditions — Osteoarthritis; Joint Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pyrocardan® implant (Active Comparator)
  Interventions: Procedure: Pyrocardan® implant
- Ligament reconstruction and tendon interposition (LRTI) (Active Comparator)
  Interventions: Procedure: Ligament reconstruction and tendon interposition (LRTI)

INTERVENTIONS:
Procedure: Pyrocardan® implant — Biconcave-shaped CMC-1 interposition implant
  Arms: Pyrocardan® implant
Procedure: Ligament reconstruction and tendon interposition (LRTI) — Weilby slightly modified as described by Burton and Pellegrini
  Arms: Ligament reconstruction and tendon interposition (LRTI)

SUMMARY:
This is a randomized controlled trial comparing the Pyrocardan® implant (intervention group) with the standard ligament reconstruction and tendon interposition (LRTI) (control group). All Danish citizens with osteoarthritis of the thumb carpometacarpal joint referred to the orthopedic department at Copenhagen University Hospital in Herlev/Gentofte will be considered for participation in the trial. The following exclude from participation in the study: Below 40 years of age; cognitive or linguistic impairment; osteoarthritis of other carpal bones; previous surgery in the carpometacarpal joint; patients with rheumatoid arthritis. A total of 64 patients will be included. The primary outcome is the patient reported outcomes questionnaire; Quick-DASH. The secondary outcomes are patient-reported outcomes, functional outcomes, radiographic outcomes, readmission, complications, revisions. The patients are examined before surgery and 3, 6, 12 and 24 months after the operation. The patients are also contacted after 5 and 10 years.

DETAILED DESCRIPTION:
The Pyrocardan® is designed by Philippe Bellemere and has been used since 2009. It is a biconcave-shaped CMC-1 interposition implant. The biconcave shape converts the CMC-1 saddle joint into a cardan-like joint. The implant is suitable for Eaton grade 2 or 3. The advantages compared to LRTI are believed to be preserved thumb length, faster recovery following surgery, increased grip and pinch strengths and less subsidence of the CMC-1 joint.

Most recently results from the Bellemere group in 2020 have shown excellent results in 103 patients 5 years following surgery. A study by Gerace et al. reported a significant improvement in pain, QuickDASH and strength, with a revision rate of 4% and a survival rate at 96% at 5 years of follow-up. A recent review from 2022 reported 97% survival rate at 4 years and an estimated survival rate of 95% at 7 years from surgery.

The purpose of this randomized study is to compare Pyrocardan® implant (intervention group 1.) with ligament reconstruction and tendon interposition (LRTI), (intervention group 2.) in patients treated with mild to moderate CMC-1 osteoarthritis. There is to our knowledge no randomized controlled trial (RCT) studies on Pyrocardan® implant.

Hypothesis Pyrocardan® can provide a faster recovery following surgery, increased grip and pinch strengths and less subsidence of the CMC-1 joint compared to LRTI.

All patients referred to the Orthopedic Surgery Department, Hand Surgery Unit at Copenhagen University Hospital in Herlev/Gentofte with CMC-1 OA with pain in the thumb base and suspected degenerative changes and indication of surgical treatment will be eligible for inclusion. The following criteria will result in exclusion from participation in the study: Age under 40, cognitive or linguistic impairment, presence of osteoarthritis in other carpal bones, previous surgery in trapeziometacarpal joint or diagnosis of rheumatoid arthritis.

A total of 64 patients will be included in the study based on a sample size calculation using the MCID of Q-DASH. This number will also account for a maximum dropout rate of 18%. The study will be a randomized clinical trial (RCT), where participants will be assigned to one of the two surgical techniques through a randomized process. Patients will be monitored to evaluate any differences between the techniques. The primary outcome measure will be the patient-reported outcome using the QuickDASH assessment. Secondary outcomes will include pain relief, questionnaires, radiographic changes, range of motion and strength (functional outcome), readmission rates, complications, and revisions. Patients will undergo examinations before the surgery and at 6 weeks, 3 months, 6 months, 12 months, and 24 months after the surgery. Additionally, patients will be contacted 5 and 10 years following the surgery for further follow-up. The study will be conducted as a single-center study and all procedures will be performed by one of three experienced hand surgeons.

ELIGIBILITY:
Inclusion Criteria:

1. Osteoarthritis of the trapeziometacarpal joint of the thumb.
2. Insufficient effect of non-surgical treatment with symptoms severe enough to justify surgical treatment.
3. ASA score 1-3, physically fit for surgery and rehabilitation

Exclusion Criteria:

1. Below 40 years of age
2. Cognitive or linguistic impairment
3. Osteoarthritis in other carpal bones (STT OA and others)
4. Previous surgical treatment in the trapeziometacarpal joint.
5. Patients with rheumatoid arthritis

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Patient-reported outcome: QuickDASH | 6 weeks, 3 months, 6 months, 1 year, 2 years, 5 years and 10 years
  Quick version of the Disability of the arm, shoulder and hand questionnaire (QuickDASH):
  0-100 p, higher score = more disability

SECONDARY OUTCOMES:
Patient-reported outcome | 6 weeks, 3 months, 6 months, 1 year, 2 years, 5 years and 10 years
  VAS (rest), VAS (activity), 0-10 p, higher score = more pain.
  Satisfaction scores: 1-5 p, higher score = more satisfied.
Strength measurements | 6 weeks, 3 months, 6 months, 1 year, 2 years
  Hand grip and Pinch (Kg)
Radiographs | 6 weeks
  Measured subsidence on radiographs
Return to occupation | 1 year
  Postoperative sick leave

CONTACTS AND LOCATIONS:
Overall Officials: Jens Joergsholm, MD, Principal Investigator — Herlev Gentofte Hospital
Locations (1):
- Herlev and Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No